CLINICAL TRIAL: NCT03799367
Title: The Feasibility of Drug Delivery to Infants During Breastfeeding (FEDD)
Brief Title: The Feasibility of Drug Delivery to Infants During Breastfeeding
Acronym: FEDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Principal Investigator, Kathryn Beardsall, University Lecturer, University of Cambridge, Cambridge University Hospitals NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 18/LO/0551
Record Dates: First submitted 2018-07-08; First posted 2019-01-10 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Medication Systems; Breast Feeding; Milk, Human; Infant, Newborn
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Drug delivery during breastfeeding — This study aims to give a vitamin B12 supplement to babies during breastfeeding. 30 mother-infant pairs will be recruited. The supplement will be placed into a nipple shield, both of which are commercially available, and the mother will breastfeed her baby as usual. Before and after the feed, we will 1) collect a small blood sample from the baby to see whether the vitamin levels in the infant have increased, 2) ask the mother to participate in two short interviews about her expectations and experiences using the Therapeutic Nipple Shield.

SUMMARY:
Parents commonly find giving medicines to babies, using oral syringes or spoons, difficult and emotionally stressful. In developing countries, additional stress arises due to hygiene difficulties and the lack of clean water. To overcome these challenges and encourage breastfeeding, we have developed the concept of a Therapeutic Nipple Shield, a delivery system that makes it possible to give medicine and nutrients to babies during breastfeeding. It consists of a silicone nipple shield that allows the release of medicine/nutrients into human milk during the feed. Presentations of a prototype to parents and staff at the Rosie Hospital was very positive, and encouraged this clinical study. This study aims to give a vitamin B12 supplement to babies during breastfeeding. The supplement will be placed into a nipple shield, both of which are commercially available, and the mother will breastfeed her baby as usual. Before and after the feed, we will 1) collect a small blood sample from the baby to see whether the vitamin levels in the infant have increased, 2) ask the mother to participate in two short interviews about her expectations and experiences using the Therapeutic Nipple Shield.

ELIGIBILITY:
Inclusion Criteria:

No known allergy or hypersensitivity against any ingredient used in the study Infant aged up to 12 months Confident breastfeeder (exclusively or non-exclusively)

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* Not confident at breastfeeding
* Infant not feeding properly
* Allergy or hypersensitivity against any ingredient of the commercially available Methylcobalamin Vitamin B12 Tablets (Just Vitamins Ltd, UK) used in the study (infant or mother)
* Medical conditions that could negatively influence swallowing, and thus breastfeeding

Ages: 7 Days to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Detection of the change in vitamin B12 concentration in the infants' blood 6-8 hours following vitamin B12 delivery from a nipple shield device during breastfeeding | Blood sampling base line and 6-8 hours post feed
  Two infant blood samples will be taken - one base line and one post intervention

SECONDARY OUTCOMES:
Qualitative assessment of impact on maternal expectation, experience and acceptability | Interviews will be conducted prior to and post interventional feed and will last about 30-50 min.
  Semi-structured interviews will be conducted before and after vitamin B12 delivery during breastfeeding

CONTACTS AND LOCATIONS:
Locations (1):
- addenbrookes Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maier T, Peirce P, Baird L, Whitehouse SL, Slater NKH, Beardsall K. Drug delivery from a solid formulation during breastfeeding-A feasibility study with mothers and infants. PLoS One. 2022 Mar 4;17(3):e0264747. doi: 10.1371/journal.pone.0264747. eCollection 2022. PMID 35245341